CLINICAL TRIAL: NCT03333447
Title: Retrospective and Prospective Observational Study of MRI Changes in Bone and Visceral Lesions of Patients With Type 1 Gaucher Disease Treated With VPRIV® (Velaglucerase Alfa)
Acronym: EIROS
Status: Completed | Type: Observational
Sponsor: CEN Biotech (Industry)
Collaborators: BioClinica, Inc. (Industry); Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C1294
Record Dates: First submitted 2017-10-26; First posted 2017-11-07 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Gaucher Disease, Type 1; MRI
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Patients of any age or gender with confirmed diagnosis of type 1 Gaucher disease, treated with VPRIV® at the beginning of the study. Patients should have one MRI data in the 5 previous years before starting VPRIV® treatment (up to 3 months after initiation of VPRIV®.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
This study with standardized reading MRIs, will provide for the first time objective and quantified data on organomegaly (liver and spleen volumes) as well as bone alteration (Bone Marrow Burden11) of French patients treated with VPRIV®. These data will help to better assess the impact of this treatment on these parameters.

The result of this study will also answer in part to the request of the French Transparency Commission (CT: Commission de Transparence) of the French National Health Authority to provide them with data of French patients treated with VPRIV®.

DETAILED DESCRIPTION:
All data entered will be used for analysis purposes and results will be submitted to inform regulatory agencies. Patient care and management is freely determined by the participating physician, in the framework of an observational study reflecting the daily medical practice. The clinical data, the results of routine clinical and laboratory testing that are part of standard medical care for patients with Gaucher disease will be collected from the medical record of the patient :

* Socio-demographic characteristics
* History of the disease and context of diagnosis
* Medical background
* MRI: abdominal and bone, as defined below
* Clinical data available in the range from 3 months before or after each MRI
* Biological data available in the range from 3 months before or after each MRI
* Treatment with VPRIV® (velaglucerase alfa), including the doses and regimens.

The MRI images collected during the study:

The MRIs performed in the patient's usual medical follow-up for its Gaucher disease (abdominal MRI (liver and spleen) and bone MRI (back injury pelvis, lower limbs) and / or whole-body MRI) will be collected. Among the MRIs available in the patient's medical records, MRIs will be collected as following:

* Reference MRI: MRI closest to the date of initiation of VPRIV® in the five years preceding the start of treatment or within three months after initiation of VPRIV®.
* MRIs of the retrospective phase of the study: All MRIs available between the reference MRI and the inclusion date of the patient.
* MRIs of the prospective phase of the study: all the MRIs that will be realized during the prospective phase of the study, that is to say during the year following the date patient inclusion in the study

Second reading of the MRI

The collected MRIs will be subject to a second reading, which will be conducted centrally by a medical image processing center (BioClinica).

This second reading of MRIs will particularly provide quantitative data not available initially in the patient records, such as Bone Marrow Burden (BMB) score at the lumbar spine and femur, and liver and spleen volumes.

In case the second reading provides additional data to the first reading, as any new comments or discordant diagnosis, the investigating doctor will integrate these data as soon as he has knowledge of them in the medical care of the patient.

MRI collection and transmission

Except the data from the second reading of MRIs by BioClinica, all data defined above, will be collected in the case report of the study, from the patient's medical record.

For the second centralized reading of the MRIs, the MRIs will be transmitted as follows: the investigation center will make a copy on Compact Disc - Read Only Memory (CD-ROM) of each MRI collected for the study needs, and will replace the identity the patient by an identification number whose correspondence with the patient's identity is only known by the investigation center. This patient identification number will be predefined and attributed to the patient's MRI when the patient is included in the study.

Copies of MRIs and coded will be sent securely at BioClinica center for analysis. In case of connection failure from the participating centers, MRI scans will be sent by post.

Data from this second reading by BioClinica will be retrieved for analysis. The results of the second reading by BioClinica will be forwarded to investigation center, which will include them in the patient's record.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any age or gender with confirmed diagnosis of type 1 Gaucher disease,
2. Patients treated with VPRIV® at the beginning of the study. Prior starting VPRIV® patients could be either treatment naïve or previously treated with any other Gaucher treatment than VPRIV®
3. Patients should have one MRI data in the 5 previous years before starting VPRIV® Treatment (up to 3 months after initiation of VPRIV®
4. Informed written consent obtained from the patient, and/or patient's parent(s), and/or legal representative. Assent, if old enough to grant, will be obtained from all patients under the age of 18 years

Exclusion Criteria:

1. Patients for whom MRI is contra-indicated
2. Patients who did not had an MRI during the five years prior to the initiation of treatment with VPRIV® or within three months after initiation of VPRIV®.
3. Patients included in an ongoing clinical trial where the product is blinded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To reflect the daily practices, this study includes all patients with a confirmed diagnosis of Type 1 Gaucher disease treated with VPRIV® at the date of beginning of the study and who meet the selection criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
The change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T1 measured at the femur. | 2 YEARS
  To describe changes in bone disease in femur in Gaucher's disease patients treated with Velaglucerase alfa measured by MRI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T1 measured at the femur.
The change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T2 measured at the femur. | 2 YEARS
  To describe changes in bone disease in femur in Gaucher's disease patients treated with Velaglucerase alfa measured by MRI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T2 measured at the femur.
The change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T1 measured at the lumbar spine. | 2 YEARS
  To describe changes in bone disease in lumbar spine in Gaucher's disease patients treated with Velaglucerase alfa measured by MRI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T1 measured at the lumbar spine.
The change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T2 measured at the lumbar spine. | 2 YEARS
  To describe changes in bone disease in lumbar spine in Gaucher's disease patients treated with Velaglucerase alfa measured by MRI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the BMB score weighted at T2 measured at the lumbar spine.

SECONDARY OUTCOMES:
Describe socio-demographic characteristics of patients : age | 2 YEARS
  To describe the socio-demographic of patients : age
Describe socio-demographic characteristics of patients : sex | 2 YEARS
  To describe the socio-demographic of patients : sex
Describe socio-demographic characteristics of patients : occupation | 2 YEARS
  To describe the socio-demographic of patients : occupation
Clinical evolution of patients :weight (kg) | 2 YEARS
  To describe the clinical evolution of patients : weight (kg)
Clinical evolution of patients : height (cm) | 2 YEARS
  To describe the clinical evolution of patients : height (cm)
Clinical evolution of patients : absence or presence (mild, moderate or severe) asthenia | 2 YEARS
  To describe the clinical evolution of patients : absence or presence (mild, moderate or severe) asthenia
Clinical evolution of patients : abdominal pain | 2 YEARS
  To describe the clinical evolution of patients : abdominal pain
Clinical evolution of patients : chronic bone pain | 2 YEARS
  To describe the clinical evolution of patients : chronic bone pain
Clinical evolution of patients : bone crises | 2 YEARS
  To describe the clinical evolution of patients : bone crises
Clinical evolution of patients : bleeding and hemorrhagic syndrome | 2 YEARS
  To describe the clinical evolution of patients : bleeding and hemorrhagic syndrome
Clinical evolution of patients : pulmonary impairment | 2 YEARS
  To describe the clinical evolution of patients : pulmonary impairment
Clinical evolution of patients : neurological impairment | 2 YEARS
  To describe the clinical evolution of patients : neurological impairment
Clinical evolution of patient : absence or presence of hepatomegaly | 2 YEARS
  To describe the clinical evolution of patients : absence or presence of hepatomegaly, with the extent of the arrow (medio-clavicular line) (cm)
Clinical evolution of patients : absence or presence of splenomegaly | 2 YEARS
  To describe the clinical evolution of patients : absence or presence of splenomegaly, with the extent of the costal overhang (cm)
Evolution of the parameters measured by MRI : Bone alterations | 2 YEARS
  To describe the evolution of the parameters measured by MRI : bone alterations (spine, pelvis, femurs, tibias and other symptomatic localization). Absence or presence of bone lesions and their locations: bone infiltration, cortical thinning, osteonecrosis, bone infarction, stroke sequelae, vertebral compression, fracture or other bone disease.
  If possible, compare the evolution of MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Liver evaluation : absence or presence of hepatomegaly with the extent of the arrow (medio-clavicular line) (cm). | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Visceral involvement : Liver evaluation criteria MRI : absence or presence of hepatomegaly, with the extent of the arrow (medio-clavicular line) (cm).
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Liver evaluation : evolution of the liver volume (m3). | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Liver evaluation criteria MRI : evolution of the liver volume (m3).
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Spleen evaluation : absence or presence of splenomegaly | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Spleen evaluation MRI : absence or presence of splenomegaly.
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Spleen evaluation : evolution of the extent of the costal overhang (cm) | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Spleen evaluation MRI : evolution of the extent of the costal overhang (cm).
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Spleen evaluation : absence or presence of splenomegaly. | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Spleen evaluation MRI : absence or presence of splenomegaly.
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Spleen evaluation : evolution of the spleen volume (m3) | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Spleen evaluation MRI : evolution of the spleen volume (m3).
  If possible, compare the evolution of this MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of the parameters measured by MRI : Presence or absence of myocardia alterations | 2 YEARS
  To describe the evolution of the parameters measured by MRI : Presence or absence of myocardial, nodules, fibrosis, vesicular stones or other alterations.
  If possible, compare the evolution of MRI parameters between treatment-naive patients and patients previously treated with another specific treatment for Gaucher disease at the baseline MRI.
Evolution of Biological parameters : hemoglobin (g/dl) | 2 YEARS
  To describe the evolution of biological parameters : hemoglobin (g/dl)
Evolution of Biological parameters : leukocytes (cells/mm3) | 2 YEARS
  To describe the evolution of biological parameters : leukocytes (cells/mm3)
Evolution of Biological parameters : platelets (mm3) | 2 YEARS
  To describe the evolution of biological parameters : platelets (mm3)
Evolution of Biological parameters : Angiotensin Converting Enzyme (ACE) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : ACE (angiotensin converting enzyme (U/l)
Evolution of Biological parameters: ferritin (mg/l) | 2 YEARS
  To describe the evolution of biological parameters : ferritin (mg/l)
Evolution of Biological parameters : chitotriosidase (nmol/h/ml) | 2 YEARS
  To describe the evolution of biological parameters : chitotriosidase (nmol/h/ml)
Evolution of Biological parameters : CCL18 (ng/ml) | 2 YEARS
  To describe the evolution of biological parameters : CCL18 (ng/ml)
Evolution of Biological parameters : vitamin D (nmol/L) | 2 YEARS
  To describe the evolution of biological parameters : vitamin D (nmol/L)
Evolution of Biological parameters : vitamin B12 (pmol/l) | 2 YEARS
  To describe the evolution of biological parameters : vitamin B12 (pmol/l)
Evolution of Biological parameters : serum glutamate oxaloacetate transaminase (SGOT) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : SGOT (U/l)
Evolution of Biological parameters : Aspartate aminotransferase (AST) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : AST (U/l)
Evolution of Biological parameters : serum glutamate pyruvate transaminase (SGPT) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : SGPT (U/l)
Evolution of Biological parameters : Alanine Aminotransferase (ALT) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : ALT (U/l)
Evolution of Biological parameters : Gamma-glutamyltransferase (GGT) (U/l) | 2 YEARS
  To describe the evolution of biological parameters : GGT (U/l)
Evolution of Biological parameters : alkaline phosphatase (U/l) | 2 YEARS
  To describe the evolution of biological parameters : alkaline phosphatase (U/l)
Evolution of Biological parameters : triglycerides (mmol/l) | 2 YEARS
  To describe the evolution of biological parameters : triglycerides (mmol/l)
Evolution of Biological parameters : total cholesterol (mmol/l) | 2 YEARS
  To describe the evolution of biological parameters : total cholesterol (mmol/l)
Evolution of Biological parameters : gamma globulin (g/l) | 2 YEARS
  To describe the evolution of biological parameters : gamma globulin (g/l).
Evolution of Biological parameters : serum calcium (mmol/l) | 2 YEARS
  To describe the evolution of biological parameters : serum calcium (mmol/l)
Evolution of Biological parameters : presence or absence of a monoclonal peak and the type if any. | 2 YEARS
  To describe the evolution of biological parameters : presence or absence of a monoclonal peak and the type if any.

CONTACTS AND LOCATIONS:
Locations (1):
- Beaujon Hospital, Clichy, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT03333447/Prot_000.pdf